CLINICAL TRIAL: NCT05868408
Title: Effect of Partially Hydrolyzed, Whey-based Infant Formulas on Growth and Tolerability in Healthy Term Infants: a Double-blind, Randomized, Controlled, Multi-arm Trial
Brief Title: Effect of Partially Hydrolyzed, Whey-based Infant Formulas on Growth and Tolerability in Healthy Term Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 21.10.INF
Record Dates: First submitted 2023-03-16; First posted 2023-05-22 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Infant Nutritional Physiological Phenomena; Infant Formula; Infant Health; Infant Development; Growth and Development

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, controlled, multi-arm trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control formula (Active Comparator): CTRL, an infant formula with minimum protein content of 1.8g intact protein/100kcal
  Interventions: Other: Control Formula
- Experimental formula 1 (Experimental): EXPL1, an infant formula with minimum protein content of 1.9g hydrolyzed protein/100kcal
  Interventions: Other: Experimental Formula 1
- Experimental formula 2 (Experimental): EXPL2, an infant formula identical to EXPL1 but manufactured using a different partially hydrolyzed milk protein base
  Interventions: Other: Experimental Formula 2

INTERVENTIONS:
Other: Control Formula — Infant formula made with intact protein - minimum 1.8g protein/100kcal
  Arms: Control formula
Other: Experimental Formula 1 — Infant formula made with hydrolyzed protein - minimum 1.9g protein/100kcal
  Arms: Experimental formula 1
Other: Experimental Formula 2 — Infant formula made with hydrolyzed protein - minimum 1.9g protein/100kcal
  Arms: Experimental formula 2

SUMMARY:
This study will assess the effect of partially hydrolyzed, whey-based infant formulas on growth and gastrointestinal tolerance in healthy term infants.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent has been obtained from at least one parent (or other legally acceptable representative [LAR]), if applicable)
2. Infant gestational age ≥37 completed weeks
3. Infant birth weight of ≥2.5 kg and ≤4.5 kg
4. Singleton birth
5. Infant postnatal age ≤28 days (date of birth = day 0)
6. Mother has previously decided to fully formula-feed, and infant is no longer breastfeeding or receiving breast milk
7. Infant's parent(s)/LAR is of legal age of majority, must understand the informed consent form and other relevant study documents, and is willing and able to fulfill the requirements of the study protocol

Exclusion Criteria:

1. Chronic infectious, metabolic, genetic illness or other disease, including any condition that impacts feeding or growth
2. Major congenital or chromosomal abnormality known to affect growth (e.g., congenital heart disease, cystic fibrosis)
3. Maternal medical conditions known to affect infant growth (e.g., untreated preeclampsia or gestational diabetes)
4. Infants with special dietary needs other than standard infant formula
5. Infants with known (or symptoms suggestive of) cow's milk protein intolerance/allergy, or lactose intolerance or severe food allergies that impact diet
6. Child has other medical or psychiatric condition that, in the judgement of the investigator, would make the child inappropriate for entry into the study
7. Currently participating or having participated in another interventional clinical trial prior to enrollment

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 234 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Difference in growth in first 4 months of life between control and experimental groups | From enrollment to age 4 months
  To demonstrate that growth from enrollment to age 4 months of infants fed experimental formula 1 (EXPL1) or experimental formula 2 (EXPL2) is non-inferior to that of infants fed control formula (CTRL). This is measured by weight gain velocity (g/day).
Equivalence in growth in first 4 months of life in experimental groups | From enrollment to age 4 months
  To demonstrate that growth from enrollment to age 4 months is equivalent between infants fed EXPL1 or EXPL2. This is measured by weight gain velocity (g/day).

SECONDARY OUTCOMES:
Gastrointestinal (GI) tolerance | Enrollment and age 4, 6, and 12 months
  GI tolerance assessed using the Infant Gastrointestinal Symptom Questionnaire (IGSQ). IGSQ scores range from 13 to 65, with lower scores indicating lower GI symptom burden.
Stooling pattern | Age 2 and 4 months
  Stool frequency and consistency assessed using a 3-day infant stool diary.
Atopic dermatitis severity | Enrollment and age 4, 6, and 12 months
  Atopic dermatitis severity assessed using the Patient Oriented Eczema Measure (POEM). POEM scores range from 0 to 28, with lower scores indicating lower atopic dermatitis severity.
Allergy-related symptoms | Enrollment and age 4, 6, and 12 months
  Allergy-related symptoms assessed using the Multi-Organ System Questionnaire for Infants (MOSQ-I). MOSQ-I scores range from 0 to 105, with lower scores indicating lower allergy-related symptom burden.
Dietary intake | Age 6 months
  Total energy and macronutrient intake calculated from food recalls / diaries
Weight | Enrollment and age 1, 2, 3, 4, and 6 months
  Weight (g)
Length | Enrollment and age 1, 2, 3, 4, and 6 months
  Length (cm)
Head circumference | Enrollment and age 1, 2, 3, 4, and 6 months
  Head circumference (cm)
Weight-for-age z-score | Enrollment and age 1, 2, 3, 4, and 6 months
  Weight-for-age z-score based on World Health Organization (WHO) and Saudi Arabian growth charts.
Weight-for-length z-score | Enrollment and age 1, 2, 3, 4, and 6 months
  Weight-for-length z-score based on World Health Organization (WHO) and Saudi Arabian growth charts.
Length-for-age z-score | Enrollment and age 1, 2, 3, 4, and 6 months
  Length-for-age z-score based on World Health Organization (WHO) and Saudi Arabian growth charts.
Head circumference-for-age z-score | Enrollment and age 1, 2, 3, 4, and 6 months
  Head circumference-for-age z-score based on World Health Organization (WHO) and Saudi Arabian growth charts.

OTHER OUTCOMES:
Stool microbiota composition | Age 4 months
  Stool microbiota composition assessed using shotgun metagenomic analysis
Stool microbiota metabolism | Age 4 months
  Stool organic acids and other metabolites
Fecal peptides | Age 4 months
  Fecal milk-derived peptides
Urinary metabolomic profile | Age 4 months
  Untargeted analysis of urine metabolites by H1-nuclear magnetic resonance (NMR) spectroscopy

CONTACTS AND LOCATIONS:
Locations (3):
- Saudi Arabia (3):
  - National Guard Hospital, Jeddah
  - King Faisal Specialist Hospital and Research Center, Riyadh
  - National Guard Hospital, Riyadh

IPD SHARING:
Plan to Share IPD: No